CLINICAL TRIAL: NCT02707913
Title: Clinical Bioequivalence Study on Two Amlodipine Tablet 10mg Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BABE-P15-097
Record Dates: First submitted 2016-03-10; First posted 2016-03-14 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BF-Amlodipine Tablet 10mg (Experimental): During the study session, healthy subjects will be administered a single dose of BF-Amlodipine Tablet 10mg after an overnight fast of approximately 10 hours
  Interventions: Drug: BF-Amlodipine Tablet 10mg
- Norvasc Tablet 10mg (Active Comparator): During the study session, healthy subjects will be administered a single dose of Norvasc Tablet 10mg after an overnight fast of approximately 10 hours
  Interventions: Drug: Norvasc Tablet 10mg

INTERVENTIONS:
Drug: BF-Amlodipine Tablet 10mg — BF-Amlodipine Tablet 10mg is a generic product manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited
  Other Names: Amlodipine Tablet 10mg
  Arms: BF-Amlodipine Tablet 10mg
Drug: Norvasc Tablet 10mg — Norvasc Tablet 10mg will be used as a comparator drug for the BE study
  Other Names: Amlodipine Tablet 10mg
  Arms: Norvasc Tablet 10mg

SUMMARY:
The purpose of the study is to compare the bioavailability of a generic product of amlodipine with that of a reference product when administered to healthy volunteers under fasting conditions. The test product name is BF-Amlodipine Tablet 10mg manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited, and the reference product is Norvasc Tablet 10mg. The plasma pharmacokinetic data of amlodipine obtained from two formulations will be used to access the interchangeability of the products

DETAILED DESCRIPTION:
The study design is a single-dose, two-treatment, two-period, two-sequence crossover with a washout period of two to three weeks. During each session, the subjects will be administered a single oral dose of 10mg amlodipine (one BF-Amlodipine Tablet 10mg or one Norvasc Tablet 10mg) after an overnight fast of approximately 10 hours. Venous blood samples will be collected at pre-dose (0 h), and up to 96 h post dose. The plasma concentrations of amlodipine will be determined by a validated assay. The non-compartmental method will be used to analyze the plasma concentration-time data and calculate the main pharmacokinetic parameters such as Peak plasma concentration (Cmax), Time to maximum concentration (Tmax), Area under the plasma concentration versus time curve (AUC0-last, AUC0-inf) and Elimination half-life (T1/2). Analysis of Variance (ANOVA) will be conducted on logarithmically transformed Cmax, AUC0-last and AUC0-inf. The two one sided tests will be used to calculate the 90% confidence intervals for the mean difference in AUC0-last, AUC0-inf and Cmax, and to assess the bioequivalence of the two products

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18 to 27
* Accessible vein for blood sampling
* High probability for compliance and completion of the study
* No significant abnormalities in general physical examination
* Electrocardiogram (ECG) recording within normal limits
* Biochemical and haematological parameters within normal limits
* Subjects must agree to take effective contraceptive methods to prevent pregnancy from the start of screening until two weeks of last dose administration

Exclusion Criteria:

* History of hepatic, renal, biliary, cardiovascular, gastrointestinal, haematological and other chronic and acute diseases within 3 months prior to the study
* Clinically relevant abnormality in physical examination, ECG evaluation, urine test, blood chemistry and haematological test
* Tobacco use in any forms
* Regular consumer of alcohol
* Blood donation within 4 weeks prior to the start of the study
* Use of amlodipine within 4 weeks before the study
* Use of antihypertensive medications within 4 weeks before the study
* Volunteer in any other clinical drug study within 2 months prior to this study
* Hypersensitivity to amlodipine or other drugs in its class
* History of drug abuse in any form
* Female subjects who are breastfeeding or pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of amlodipine | 96 hours
Area under the plasma concentration versus time curve (AUC) of amlodipine | 96 hours

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of amlodipine | 96 hours
Elimination half-life (t1/2) of amlodipine) | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zhong ZUO, Principal Investigator — School of Pharmacy, The Chinese Univesity of Hong Kong; Risa Ozaki, Study Director — Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong; Brian Tomlinson, Study Director — Dept. of Medicine and Therapeutics, The Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
Study investigators and his/her study team members, domestic and foreign regulatory agencies, the Institutional Review Board/Ethics Committee (IRB/EC) involved in the study, and laboratories and other individuals and organizations that analyze the subjects' protected health information in connection with this study have access to the data or study